CLINICAL TRIAL: NCT05097235
Title: Type III PROGRESS Framework for Prognosis Research: Building Prognostic Models for Sensory Profiles in the Development of Central Sensitisation in the Chronic Low Back Pain Population
Brief Title: Type 3 Predictive Observational Study for Sensory Profiles in Central Sensitization in Low Back Pain Population.
Acronym: T3PredCohSt
Status: Completed | Type: Observational
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Pieter Graper, Principal Investigator, Vrije Universiteit Brussel
Other Study IDs: T-3LoCoSt
Record Dates: First submitted 2021-10-13; First posted 2021-10-28 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Sensory Profiles, Nociplastic Pain, Low Back Pain
Keywords: sensory profiles, central sensitization, low back pain.
MeSH Terms: conditions — Nociplastic Pain; Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- t0, t1: acute low back pain, inclusion criteria.

SUMMARY:
This study conducts prognostic research to develop, validate, and evaluate the predictive role of sensory profiles in the development of sensory profiles over time. Therefore, a type 3 prognostic model research will be conducted in the low back pain population.

DETAILED DESCRIPTION:
This is a longitudinal multi-centre prospective cohort study design with two measurements.The STROBE statement is used as guideline and the results are reported according to the TRIPOD, and REMARK checklists. The study is a type III prognostic model research study, following the PROGRESS framework to assess the outcome by the development, validation, and evaluation of the impact of incorporating single or multiple prognostic factors, and their prognostic value at baseline in the development of CS over a period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute LBP (< six weeks)
* with or without radiating pain
* aged 18 to 60 years
* a pain-free episode for at least 12 weeks before the onset of their current back pain.
* be able to read and understand the Dutch language.

Exclusion Criteria:

* any specific cause of low back pain

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: -primary physiotherapy practices in the Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Central Sensitization Inventory | 12 weeks
  Central Sensitization Inventory (CSI) is a questionnaire which consists of 2 parts. Part A measures 25 symptoms on a 5-point scale, scoring ranges from 0-4, with a total on an ordinal scale ranging from 0-100. Part B records the presence diagnosed central sensitization syndromes, on a nominal scale. Four factors with excellent internal consistency (Cronbach's alpha= 0.91) can be identified: disability and physical symptoms; higher central sensitivity; urological and dermatological symptoms and emotional distress. The CSI has an excellent test-retest reliability of ICC=0.88 in chronic low back pain populations.

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Scafoglieri, PhD, Principal Investigator — Vrije Universiteit Brussel, Brussels, Belgium
Locations (1):
- Fysiomobilae, Zwolle, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No